CLINICAL TRIAL: NCT00683943
Title: Pilot Study of Tolerability of Lithium Therapy in Patients With Spinocerebellar Ataxia Type I (SCA1)
Brief Title: Lithium Treatment for Patients With Spinocerebellar Ataxia Type I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080134; 08-N-0134
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-02-27

CONDITIONS: Spinocerebellar Ataxia Type I
Keywords: Spinocerebellar Ataxia; Lithium
MeSH Terms: conditions — Spinocerebellar Ataxias | interventions — Lithium Carbonate

INTERVENTIONS:
Drug: Lithium Carbonate

SUMMARY:
This study will evaluate the side effects and tolerability of the drug lithium in patients with spinocerebellar ataxia type I (SCA1) an inherited disorder caused by loss of nerve cells in parts of the brain. Symptoms include ataxia (difficulty walking) and loss of muscle coordination and strength. Recent studies suggest that lithium may be helpful in treating some SCA1 symptoms.

People between 18 and 65 years of age with SCA1 who have only difficulty walking or who have difficulty walking as well as tremor, hand incoordination or speech problems, may be eligible for this study. Participation requires three hospital admissions at the NIH Clinical Center and one outpatient visit.

Participants undergo the following tests and procedures:

Admission 1 (2-6 weeks)

* Medical history, physical examination, blood and urine tests, electrocardiogram.
* Evaluation of SCA1 symptoms (balance, walking, dexterity, tremor, memory, mood and concentration).
* Monitoring of liquid intake and output (urine) and weight changes.
* Lithium treatment Start treatment and remain in hospital until the blood level of the drug is stabilized; continue treatment at home after hospital discharge.

Admission 2 (2-4 days, 4 weeks after hospital discharge).

* Repeat of some or all of the procedures done at the first admission.
* Continue lithium in hospital and at home after discharge, with local physician checking laboratory values as needed.

Admission 3 (2-4 days, 8 weeks after Admission 2).

* Repeat of some or all of the procedures done at other admissions.
* Stop lithium.

Outpatient Visit (4 weeks after Admission 3)

* Evaluation of SCA1 symptoms.
* Blood and urine tests.

DETAILED DESCRIPTION:
Objective

Evaluation of tolerability and safety of lithium in SCA1 patients.

Study Population

A total of 10 molecularly diagnosed SCA1 patients divided in two groups. One group would be composed of 5 patients with gait difficulty only and 5 patients with gait difficulty and tremor, hand incoordination or speech difficulties.

Design

Patients will be admitted to the NIH Clinical Center for initiation and titration of Lithium until high therapeutic levels currently accepted for the treatment of Bipolar affective disorder are achieved (1.0-1.2 mmol/L) or a maximum tolerated dose. During their admissions, they will have neurological evaluations, ataxia and tremor evaluations, timed-up-and-go testing, quality of life assessment, questionnaires evaluating sleep, balance confidence and depression, memory testing, alertness assessment and quantitative balance/sway evaluations. Parameters and side effect profiles will be assessed at baseline, 1 month (plus or minus 5 days) and 3 months (plus or minus 5 days) after achievement of therapeutic levels. They will also have an exit evaluation one month (plus or minus 5 days) after discontinuation of Lithium also at the NIH. For their baseline evaluation and titration, patients will be admitted to the NIH for 4 weeks plus or minus 2 weeks. Evaluation at 1 month (plus or minus 5 days) and 3 months (plus or minus 5 days)

Outcome Measures

Primary Outcomes

1. Incidence of side effects
2. Side effect profile

Secondary Outcomes

1. Timed-up-and-go test
2. ICARS score
3. SARA score
4. Modified Falls Efficacy Scale
5. Quantitative Sway/Balance assessment
6. Tremor Rating Scale:

   * Part A Tremor location/severity rating
   * Part B Handwriting and drawings
   * Part C Functional disabilities resulting from tremor
7. Questionnaires related to sleep, depression (Beck Depression Inventory) (BDI), alertness (Computerized Continuous Performing Tasks) and memory (Mini Mental State Examination)
8. Dexterity evaluation At-Home Testing Program device

ELIGIBILITY:
* INCLUSION CRITERIA:
* 18-65 years of age
* Molecularly diagnosed SCA1
* Gait disturbance only or gait disturbance and tremor and/or hand incoordination and/or speech difficulty.
* Women of childbearing age who agree to use contraceptive methods for the duration of the study.

EXCLUSION CRITERIA:

* Children
* Pregnant or nursing women
* Anyone on a low-sodium diet
* Cognitively impaired individuals
* Schizophrenics
* Family history of thyroid diseases
* Patients with medical conditions that can be affected by Lithium such as diabetes mellitus, difficulty urinating, infections (severe occurring with fever, prolonged sweating, diarrhea, or vomiting), kidney disease, epilepsy, thyroid disease, heart disease, pulmonary disease, bipolar affective disorder, cardiac arrhythmia, diabetes insipidus, Parkinson disease, psoriasis and leukemia.
* Anyone taking the following medications: diuretics, nonsteroidal anti-inflammatory agents, methyldopa, tetracycline, antipsychotic, neuromuscular blocking agents, digoxin, phenytoin, acetazolamide, calcium iodide, iodinated glycerol, potassium iodide, calcium channel blockers and/or metronidazole. Patients on these medications may be enrolled and their lithium levels will be followed very closely. If levels are consistently maintained, the subject may remain in the study.
* Age greater than 65 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-05-18; Primary Completion 2010-02-25 (Actual); Study Completion 2010-02-25 (Actual)

PRIMARY OUTCOMES:
Incidence of side effects, side effect profile, and number of falls.

SECONDARY OUTCOMES:
ICARS scores, SARA scores, Quantitative Sway/Balance assessment, Tremor Rating Scale scores, dexterity evaluation, sleep questionnaire, Computerized Continuous Performing Tasks assessment

CONTACTS AND LOCATIONS:
Overall Officials: Grisel J Lopez, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Allagui MS, Vincent C, El feki A, Gaubin Y, Croute F. Lithium toxicity and expression of stress-related genes or proteins in A549 cells. Biochim Biophys Acta. 2007 Jul;1773(7):1107-15. doi: 10.1016/j.bbamcr.2007.04.007. Epub 2007 Apr 21. PMID 17512992
- [Background] Cummings CJ, Sun Y, Opal P, Antalffy B, Mestril R, Orr HT, Dillmann WH, Zoghbi HY. Over-expression of inducible HSP70 chaperone suppresses neuropathology and improves motor function in SCA1 mice. Hum Mol Genet. 2001 Jul 1;10(14):1511-8. doi: 10.1093/hmg/10.14.1511. PMID 11448943
- [Background] de Chiara C, Menon RP, Dal Piaz F, Calder L, Pastore A. Polyglutamine is not all: the functional role of the AXH domain in the ataxin-1 protein. J Mol Biol. 2005 Dec 9;354(4):883-93. doi: 10.1016/j.jmb.2005.09.083. Epub 2005 Oct 18. PMID 16277991